CLINICAL TRIAL: NCT06900426
Title: Lung Atelectasis Improvement Through Positive End Expiratory Pressure During Anesthetic Induction: a Randomized Trial
Brief Title: Lung Atelectasis Improvement Through Positive End Expiratory Pressure During Anesthetic Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jun Zhang, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2502-Exp148
Record Dates: First submitted 2025-03-17; First posted 2025-03-28 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Lung Injury, Acute
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PEEP0 (Other): There is ZEEP during anesthetic induction
  Interventions: Other: ZEEP
- PEEP5 (Experimental): There is 5 cmH2O PEEP during anesthetic induction.
  Interventions: Other: 5PEEP
- PEEP10 (Experimental): There is 10 cmH2O PEEP during anesthetic induction.
  Interventions: Other: 10 PEEP

INTERVENTIONS:
Other: 10 PEEP — Using 10cmH2O PEEP during anesthetic induction monitored by EIT.
  Arms: PEEP10
Other: ZEEP — No PEEP
  Arms: PEEP0
Other: 5PEEP — Using 5cmH2O PEEP
  Arms: PEEP5

SUMMARY:
Anesthetic induction could lead to lung atelectasis, increase intrapulmonary shunt, and potentially impair oxygenation. The study aimed to validate that a positive end-expiratory pressure (PEEP) of 10 cmH2O could reduce lung atelectasis, comparing to 0 or 5 cmH2O with limited overdistension.

DETAILED DESCRIPTION:
General anesthesia may introduce lung atelectasis, which causes an increase in intrapulmonary shunt, and impairs oxygenation, even in the lung-healthy subjects. The magnitude of shunt is correlated with the formation of pulmonary atelectasis. The study aimed to validate that a positive end-expiratory pressure (PEEP) of 10 cmH2O could reduce lung atelectasis, comparing to 0 or 5 cmH2O with limited overdistension. Surgical patients with healthy lungs were randomly assigned to receive 0, 5 or 10 cmH2O PEEP (PEEP0, PEEP5 and PEEP10 groups). Anesthetic induction was performed by certified registered anesthesiologists, during which the patients were mechanically ventilated using the volume-controlled mode. Electrical impedance tomography (EIT) was used to dynamically assess the lung atelectasis during anesthetic induction (spontaneous, mask, and endotracheal intubation ventilation). The primary outcome was the dorsal change of end expiratory lung impedance (△EELI) after 2 mins anesthetic induction. The secondary outcome was driving pressure, EIT-derived ventilation homogeneity, hemodynamics and PaO2/FiO2.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 80 years
* scheduled for elective non-cardiothoracic cancer surgery
* general anesthesia.

Exclusion Criteria:

* acute or chronic respiratory disorders, such as chronic obstructive pulmonary disease (COPD) or asthma;
* a history of lung surgery
* a high risk of reflux and aspiration
* a requirement for awake intubation
* facial or thoracic deformities
* the presence of implants, such as cardiac pacemakers
* pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
the dorsal △EELV after 2 minutes anesthetic induction | 2 minutes after anesthetic induction
  The primary outcome was the dorsal △EELV after 2 minutes anesthetic induction (endotracheal intubation ventilation) monitored by EIT.

SECONDARY OUTCOMES:
driving pressure | 2 minutes after anesthetic induction
  Pplat - PEEP
GI | 2 minutes after anesthetic induction
  Global imhomogeneity monitored by EIT
CoV | 2 minutes after anesthetic induction
  The central of ventilation monitored by EIT
hemodynamics | During anesthetic induction
  Blood pressure
PaO2/FiO2 | During anesthetic induction
  PaO2/FiO2 during anesthetic induction

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Professor, Principal Investigator — Fudan University Shanghai Cancer Centre
Locations (1):
- Fudan University Shanghai Cancer Centre, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data sets are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start date：The study was officially published. End date：Two years after the study was officially published.
Access Criteria: The data sets are available from the corresponding author through email on reasonable request by reletive investigators.